CLINICAL TRIAL: NCT04169074
Title: Immune Modulation by Abemaciclib in HPV-Negative Head and Neck Squamous Cell Carcinoma (HNSCC): A Phase II Window Trial.
Brief Title: Immune Modulation by Abemaciclib in Head and Neck Squamous Cell Carcinoma (HNSCC). (AIM Trial)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Standard of care therapy for Stage III-IVA HNSCC updated in June to include neoadjuvant + adjuvant immunotherapy.
Sponsor: University of Arizona (Other)
Collaborators: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1906702171
Record Dates: First submitted 2019-04-15; First posted 2019-11-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: HNSCC
Keywords: Head and Neck Cancer; HNSCC; Squamous Cell Cancer; abemaciclib
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Neoplasms, Squamous Cell | interventions — abemaciclib

STUDY DESIGN:
Intervention Model Description: This is an open label Phase II single-arm window trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with abemaciclib (Experimental): Treatment will consist of a single neoadjuvant cycle of 10-21 days (+7 days if needed due to surgical delay). Abemaciclib will be administered from days 1-21. Abemaciclib may be continued for an additional 7 days, or up to 28 days, for delays in planned surgery. Abemaciclib 200 mg PO twice daily on Days 1-21 (+7 days).
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Treatment will consist of a single neoadjuvant cycle of 10-21 days (+7 days). Abemaciclib will be administered from days 1-21. Abemaciclib may be continued for an additional 7 days, or up to 28 days, for delays in planned surgery.

SUMMARY:
This is a Phase II single-arm window trial to assess the clinical and biological effects of neoadjuvant abemaciclib in patients with HPV-negative head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
This is a Phase II single-arm window trial to assess the clinical and biological effects of 10-21 days of neoadjuvant abemaciclib in patients with HPV-negative HNSCC who are planned for oncologic surgery, with pre-clinically informed genetic and immune biomarker correlatives.

In the window-of-opportunity clinical trial, patients planned for oncologic surgery are briefly exposed to a novel cancer agent in the window between diagnostic biopsy and definitive surgery. Paired, pre- and post-surgical tumor specimens permit ex vivo analysis of target modulation in both tumor and the tumor microenvironment - providing insight into mechanism of action and paving the way for rigorous companion biomarker development. Clinical activity is assessed by quantitative change in tumor size (∆T), which is correlated to hypothesis-driven genomic and immune biomarkers of interest.

Investigators hypothesize that abemaciclib will significantly reduce tumor burden as measured by ∆T. Further, investigators will test the primary biomarker hypothesis that the clinical activity of abemaciclib is associated with an increased proportion of tumors that are T-cell inflamed. Investigators will evaluate tumor-intrinsic, tumor microenvironment (TME), and microbiome biomarker hypotheses in specific genetic contexts, including tumors with specific classes of tumor protein 53 (TP53) mutations, p16 loss, and/or CCND1 amplification.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or histologic diagnosis of squamous cell carcinoma of the oral cavity, p16-negative oropharynx, hypopharynx, or larynx.
2. Tumors must be HPV-negative. For eligibility, tumors of the oral cavity, hypopharynx, or larynx will be considered HPV-negative without specialized testing. Tumors of the oropharynx must be HPV-negative as determined by p16 immunohistochemistry and/or HPV-DNA per local standard.
3. Clinical stage I-IVa based upon the American Joint Committee on Cancer (AJCC) staging manual, 8th edition.
4. Appropriate and planned for oncologic resection of the primary tumor and/or neck dissection.
5. Clinically or radiologically measurable disease; the primary tumor and/or cervical nodes may be measurable according to RECIST 1.1 (tumor diameter ≥ 1 cm; short-axis lymph node diameter ≥ 1.5 cm) OR by caliper/ruler measurement (tumor diameter ≥ 1 cm).
6. No prior treatment for the index (study-qualifying) HNSCC.
7. Patients with two simultaneous primary tumors or bilateral tumors are included.
8. The index HNSCC may be a second primary HNSCC, provided the following criteria are met:

   a. The previously treated HNSCC was treated with curative intent. b. The index HNSCC is at least 1 cm from the previously treated HNSCC. c. At least 2 years have elapsed since curative treatment of the previous HNSCC without evidence for recurrence.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1. (See Appendix 1.)
10. Adequate hematologic function, as defined by:

    a. Absolute neutrophil count (ANC) ≥ 1,500/µl b. Platelets ≥ 100,000/µl c. Hemoglobin ≥ 8 g/dL
11. Adequate liver function, as defined by:

    a. Bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). Patients with Gilbert's syndrome with a total bilirubin ≤ 2.0 x ULN and direct bilirubin within normal limits are permitted.

    b. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN
12. Adequate renal function, as defined by creatinine ≤ 1.5 x ULN.
13. Able to swallow oral medications.
14. Have signed written informed consent.
15. Consent to biomarker collection requirements, including mandatory baseline and intra-operative research biopsies of the index tumor.

Exclusion Criteria:

1. Prior treatment with any cyclin-dependent kinase (CDK) 4/6 inhibitor or anti-programmed death (PD)-1/L1 inhibitor is not allowed.
2. Current or prior use of immunosuppressive medication within 14 days before the first dose of their assigned protocol treatment. The following are exceptions to this criterion unless otherwise indicated:

   1. Intranasal, inhaled, or topical steroids, or local steroid injections (eg, intra articular injection)
   2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   3. Steroids as premedication for hypersensitivity reactions (eg, CT premedication) and/or as anti-emetics
3. Active or previously documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis, Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement. Subclinical hypothyroidism (eg. Elevated thyroid-stimulating hormone (TSH), low or normal free T4, and asymptomatic) observed on screening labs is not an exclusion.
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study PI
   5. Patients with celiac disease controlled by diet alone
4. Patient has a personal history of any of the following cardiac or pulmonary abnormalities:

   1. Syncope of cardiovascular etiology
   2. Ventricular arrhythmia of pathologic origin (including, but limited to, ventricular tachycardia and ventricular fibrillation)
   3. Sudden cardiac arrest
   4. Documented history of New York Heart Association functional classification III-IV congestive heart failure
   5. Myocardial infarction ≤ 6 months prior to enrollment
   6. Current unstable angina pectoris
   7. Interstitial lung disease
   8. Severe dyspnea at rest or requiring oxygen therapy
5. Patient with impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral abemaciclib (e.g. history of major surgical resection involving the stomach or small bowel, malabsorption syndrome, preexisting Crohn's disease or ulcerative colitis, preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
6. Patients who require the chronic administration of drugs that are strong and moderate inducers of Cytochrome P450, family 3, subfamily A, (CYP3A) and/or strong inhibitors of CYP3A, and no acceptable substitute can be identified, are not eligible for study (See Appendix 2). Such drugs should be discontinued at least 7 days before the start of study treatment.
7. The patient has active bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or known active hepatitis B or C [e.g. hepatitis B surface antigen positive or hepatitis C antibody positive with detectable viral load]). Screening for HIV or hepatitis is not required for enrollment.
8. Patient with any other condition that would, in the Investigator's judgment, preclude patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. social/psychological complications.
9. Pregnant or nursing (lactating) women.
10. Patient who does not apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment:

    1. Sexually active males should use a condom during intercourse while taking abemaciclib and for 4 weeks after the final dose of abemaciclib.
    2. Males who are sexually active with a woman of child-bearing potential should apply highly effective contraception during the study as defined below, in order not to father a child in this period.
    3. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through at least 3 weeks after the final dose of abemaciclib. Highly effective contraception is defined as:

    i. Total abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception].

ii. Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment.

iii. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female study subjects, the vasectomized male partner should be the sole partner for that patient.] iv. Use a combination of the following (both 1+2):

1. Placement of an intrauterine device (IUD) or intrauterine system (IUS) 2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

v. Note: Hormonal contraception methods (e.g. oral, injected, and implanted) are not allowed as abemaciclib may decrease the effectiveness of hormonal contraceptives.

vi. Note: Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago.

11. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Measure quantitative change in tumor size to assess the clinical activity of abemaciclib. | Two months
  To evaluate the clinical activity of abemaciclib in patients with operable, HPV-negative HNSCC as measured by quantitative change in tumor size (∆T)1 following 10-21 (+7) days of neoadjuvant exposure. This will be measured using established RECIST v1.1 metrics for index lesions. Index lesions will be evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumor (RECIST) Committee 71.

SECONDARY OUTCOMES:
Describe the safety and tolerability of neoadjuvant exposure to abemaciclib in accordance with NCI Common Terminology Criteria for Adverse Events (CTCAE) v.5. | Two months
  To describe the safety and tolerability of neoadjuvant exposure to abemaciclib in accordance with NCI Common Terminology Criteria for Adverse Events (CTCAE) v.5.

OTHER OUTCOMES:
Measure Interferon gamma (IFN-ɣ) gene expression signature in baseline and post-treatment tumor biopsies. | Two months
  Evaluate baseline and pharmacodynamic biomarkers within the TME associated with ∆T, including IFN-ɣ gene expression signature in baseline and post-treatment tumor biopsies. The primary biomarker hypothesis is that abemaciclib will increase the proportion of tumors that are T-cell inflamed.
Measure tumor-intrinsic genetic biomarkers utilizing tumor specimen. | Two months
  Evaluate tumor-intrinsic genetic biomarkers associated with ∆T, including somatic genetic or epigenetic alterations in CCND1, CDKN2A, and TP53 utilizing tumor specimen obtained during planned oncologic head and neck cancer surgery.
Measure the distribution of tumor-infiltrating immune cell subtypes and their activation status, as measured by nanostring. | Two months
  Evaluate baseline and pharmacodynamic biomarkers within the TME associated with ∆T, including The distribution of tumor-infiltrating immune cell subtypes and their activation status, including lymphocytes and myeloid-derived stem cells, as measured by nanostring.
Measure the distribution of tumor-infiltrating immune cell subtypes and their activation status, as measured by immunohistochemistry (IHC). | Two months
  Evaluate baseline and pharmacodynamic biomarkers within the TME associated with ∆T, including The distribution of tumor-infiltrating immune cell subtypes and their activation status, including lymphocytes and myeloid-derived stem cells, as measured by immunohistochemistry (IHC).
Measure the distribution of tumor-infiltrating immune cell subtypes and their activation status, as measured by flow cytometry. | Two months
  Evaluate baseline and pharmacodynamic biomarkers within the TME associated with ∆T, including The distribution of tumor-infiltrating immune cell subtypes and their activation status, including lymphocytes and myeloid-derived stem cells, as measured by flow cytometry.
Measure the distribution of peripheral immune cell subtypes and their activation status | Two months
  To evaluate the distribution of peripheral immune cell subtypes and their activation status, and how this is altered by abemaciclib.
Measure how serum Th1 and Th2 cytokine profiles are altered by abemaciclib. | Two months
  To evaluate serum Th1 and Th2 cytokine profiles, and how they are altered by abemaciclib.
Measure tumor-intrinsic molecular mediators of response and resistance to abemaciclib. | Two months
  Evaluate tumor-intrinsic molecular mediators of response and resistance to abemaciclib in baseline and post-treatment tumor biopsies, including expression of CDKN2A (p16), CCND1 (cyclin D1), and retinoblastoma tumor suppressor protein (pRB) retinoblastoma.
Measure change in the proliferative index (∆Ki67) in pre- and post-treatment tumor specimens. | Two months
  Evaluate the anti-proliferative activity of abemaciclib as measured by change in the proliferative index (∆Ki67) in pre- and post-treatment tumor specimens.
Describe features of the oral and intestinal microbiomes that are associated with the clinical activity of abemaciclib. | Two months
  To describe features of the oral and intestinal microbiomes that are associated with the clinical activity of abemaciclib.

CONTACTS AND LOCATIONS:
Overall Officials: Ricklie Julian, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - George Washington Cancer Center, Washington D.C., District of Columbia